CLINICAL TRIAL: NCT06385301
Title: Exercise Performance on Ambient Air vs. Commonly Prescribed Nasal Low Oxygen Therapy - a Non-Inferiority Trial in Patients With Exercise Induced Desaturation Due to Chronic Lung Diseases
Brief Title: Exercise Performance on Ambient Air vs. Low-Flow Oxygen Therapy With Chronic Lung Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Lung_disease_6MWD_SOT
Record Dates: First submitted 2024-04-17; First posted 2024-04-26 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Lung Disease Chronic; Lung Diseases, Interstitial; Lung Diseases, Obstructive
Keywords: Supplemental Oxygen Therapy; 6 Minute Walking Distance; Chronic lung diseases
MeSH Terms: conditions — Lung Diseases, Interstitial; Lung Diseases, Obstructive

STUDY DESIGN:
Intervention Model Description: Each participant is its own control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambient air (Experimental): Patient will perform tests at University Hospital Zurich on ambient air
  Interventions: Other: 6-minute walk distance (6MWD) test on ambient air
- SOT via basal cannula (Active Comparator): Supplemental Oxygen Therapy (SOT) will be provided via nasal cannula from a small oxygen concentrator while the patient performs tests at University Hospital Zurich.
  Interventions: Other: 6-minute walk distance test with supplemental oxygen (approximately 3l/min, nasal)

INTERVENTIONS:
Other: 6-minute walk distance (6MWD) test on ambient air — 6-minute walk distance (6MWD) test will be performed on ambient air according to clinical standards
  Arms: Ambient air
Other: 6-minute walk distance test with supplemental oxygen (approximately 3l/min, nasal) — 6-minute walk distance (6MWD) test will be performed according to clinical standards additionally with supplemental oxygen therapy (approximately 3l/min, nasal)
  Arms: SOT via basal cannula

SUMMARY:
The investigators aim to study the effect of SOT in subjects with chronic lung disease in submaximal exercise.

DETAILED DESCRIPTION:
Participants with lung disease who live in Switzerland will have 6-minute walk distance (6MWD) test with and without SOT at approximately 3l/min via nasal cannula according to a randomized cross-over design.

The trial aims to test that the 6MWD with SOT is non-inferior to a 6MWD in the same participant under ambient air.

Our effect size was estimated with a difference of less or equal to 35m compared under SOT compared to ambient air.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years of age
* Written informed consent
* Patients with diagnosed chronic lung disease
* Former desaturation under exercise defined as Spo2-decrease >3%- Page 3 of 4
* Treated with a stable drug therapy (with no changes for at least 14 days prior to screening)

Exclusion Criteria:

* Severe hypoxemia needing supplemental oxygen therapy defined as (partial pressure of Oxygen (PaO2) < 6.9 KiloPascal (kPa)
* Pregnancy
* Unability or contraindications to undergo the investigated intervention
* Unability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
6-minute walk distance (6MWD) with supplemental oxygen therapy (SOT) vs. ambient air | after 6 minutes
  Change in 6MWD in meter between SOT via nasal cannula vs. ambient air

SECONDARY OUTCOMES:
SpO2 at rest and peak 6MWD with SOT vs. ambient air | after 6 minutes
  Change of the arterial oxygen saturation by pulse oximetry (SpO2) at rest and at peak 6MWD with SOT vs. ambient air
Heart rate at rest and peak 6MWD with SOT vs. ambient air | after 6 minutes
  Change of heart rate (bpm) at rest and at peak 6MWD with SOT vs. ambient air
Borg dyspnea scale at rest and peak 6MWD with SOT vs. ambient air | 6 minutes
  Change of Borg dyspnea scale at rest and at peak 6MWD with SOT vs. ambient air
Borg leg fatigue scale at rest and peak 6MWD with SOT vs. ambient air | after 6 minutes
  Change of Borg leg fatigue scale at rest and at peak 6MWD with SOT vs. ambient air
Blood pressure at rest and peak 6MWD with SOT vs. ambient air | after 6 minutes
  Change of Blood pressure (mmHg) at rest and at peak 6MWD with SOT vs. ambient air

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, Prof. Dr., Principal Investigator — University Hospital Zurich, Department of Pulmonology
Locations (1):
- University Hospital Zürich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data will be provided upon request and based on a clear intention reviewed by an ethical review board